CLINICAL TRIAL: NCT05650827
Title: Feasibility and Effect of Resistance Training and Protein Supplementation in Patients With Advanced Gastroesophageal Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Rikke Krabek, MD, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18.10.22
Record Dates: First submitted 2022-12-02; First posted 2022-12-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Gastro-esophageal Cancer
Keywords: Exercise oncology; Resistance exercise; Cancer; Cancer cachexia; Protein supplements; Sarcopenia; Palliative chemotherapy
MeSH Terms: conditions — Neoplasms; Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Control (No Intervention): Participants allocated to control receive first line chemotherapy the standard patient care program, as provided by Rigshospitalet, Copenhagen, Denmark.
  Participants allocated to control are allowed to exercise on their own initiative or participate in any standard care hospital- or municipality-based exercise training program. There will be no diet restrictions.
- Exercise and protein supplements intervention group (Experimental): Participants allocated to intervention receive first line chemotherapy and the standard patient care program, as provided by Rigshospitalet, Copenhagen, Denmark.
  The intervention consists of resistance training and a daily protein supplement.
  Interventions: Behavioral: Resistance training; Dietary Supplement: Protein supplement

INTERVENTIONS:
Behavioral: Resistance training — 10 weeks of resistance training 3 times pr. week.
  Arms: Exercise and protein supplements intervention group
Dietary Supplement: Protein supplement — A daily supplement of protein to ensure a daily intake of 1,6g protein/kg bodyweight
  Arms: Exercise and protein supplements intervention group

SUMMARY:
Patients with advanced gastroesophageal cancer are in great risk of losing skeletal muscle mass and developing cancer cachexia. Low skeletal muscle mass has a negative impact on quality of life, impairs physical function, increases toxicity from anti-neoplastic treatment, as well as increases risk of death.

Resistance training and protein supplements have the potential to stimulate muscle anabolism and counteract loss of skeletal muscle mass. Therefore, the investigators have designed a randomized controlled feasibility trial to evaluate the feasibility, safety and the therapeutic effect of resistance training and protein supplements in patients with advanced gastroesophageal cancer undergoing first line chemotherapy.

A total of 54 patients with advanced gastroesophageal cancer will be recruited from the Department of Oncology, Copenhagen University Hospital, Rigshospitalet and randomly allocated 2:1 to standard care plus resistance training 3 times pr. week and a daily supplement of protein or to standard care alone.

ELIGIBILITY:
Inclusion Criteria:

* histologically verified, non-resectable cancer of the esophagus, stomach, or gastroesophageal junction
* referred to first line chemotherapy.

Exclusion Criteria:

* Age < 18
* Living outside the greater Copenhagen area
* Any other malignancy requiring active treatment
* Not eligible for chemotherapy
* Performance status > 2
* Not able to swallow liquids
* Parenteral nutrition or enteral nutrition via feeding tube
* Physical or mental disabilities that prohibit execution of test or training procedures
* Pregnancy
* Inability to understand the Danish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Exercise feasibility: Exercise sessions attendance | From baseline until end of intervention (10 weeks)
  The number of attended exercise training sessions relative to the number of planed exercise sessions
Exercise feasibility: Relative dose-intensity of protein supplement | From baseline until end of intervention (10 weeks)
  The actual amount consumed relative to the amount prescribed over the intervention period
Incidence of Serious Adverse Events (SAEs). | Baseline until end of intervention (10 weeks)
  SAE will be recorded during trial assessment visits and through medical records. This procedure will concern any SAE during the trial period. For each trial visit we will collect patients' self-report of SAEs, which may have occurred during the period since the last trial visit.

SECONDARY OUTCOMES:
Exercise feasibility: Relative dose intensity of exercise | Baseline until end of intervention (10 weeks)
  The actual dose relative to the prescribed minimum dose
Exercise feasibility: Early termination of exercise sessions | Baseline until end of intervention (10 weeks)
  Termination of an exercise session before the prescribed exercises have been performed
Exercise feasibility: Exercise intervention interruptions | Baseline until end of intervention (10 weeks)
  Incidence of exercise intervention disruptions, defined as a period of ≥ 7 days without an attended exercise session
Exercise feasibility: Permanent discontinuation | Baseline until end of intervention (10 weeks)
  Incidence of permanent withdrawal from the intervention before intervention period has ended.
Body composition and anthropometrics: Total lean mass | Baseline, end of week 10
  Changes in total lean mass, assessed by dual energy x-ray absorptiometry (DXA)
Body composition and anthropometrics: Appendicular lean mass | Baseline, end of week 10
  Changes in appendicular lean mass, assessed by DXA
Body composition and anthropometrics: Total fat mass | Baseline, end of week 10
  Changes in total fat mass, assessed by DXA
Body composition and anthropometrics: Fat percentage | Baseline, end of week 10
  Changes in fat percentage, assessed by DXA
Body composition and anthropometrics: Bone mineral density | Baseline, end of week 10
  Changes in bone mineral density, assessed by DXA
Body composition and anthropometrics: Muscle thickness | Baseline, end of week 10
  Changes in thickness of the vastus lateralis, assessed by ultrasound
Body composition and anthropometrics: Skeletal muscle index | At diagnose, after 10 weeks intervention and at 1 year follow up
  Changes in skeletal muscle index, assessed by diagnostic CT scans
Body composition and anthropometrics: Skeletal muscle attenuation | At diagnose, end of week 10
  Changes in skeletal muscle attenuation, assessed by diagnostic CT scans
Body composition and anthropometrics: Adipose tissue index | At diagnose, end of week 10
  Changes in adipose tissue index, assessed by diagnostic CT scans
Body composition and anthropometrics: Body mass | Baseline, end of week 10
  Changes in body mass
Body composition and anthropometrics: Body mass index | Baseline, end of week 10
  Changes in body mass index
Body composition and anthropometrics: Hip circumference | Baseline, end of week 10
  Changes in hip circumference
Body composition and anthropometrics: Waist circumference | Baseline, end of week 10
  Changes in waist circumference
Muscle strength: Leg press maximal muscle strenght | Baseline, end of week 10
  Changes in leg press one repetition maximum (1RM)
Muscle strength: Chest press maximal muscle strenght | Baseline, end of week 10
  Changes in chest press 1RM
Muscle strength: Hand grip strenght | Baseline, end of week 10
  Changes in hand grip strength, assessed using a dynamometer
Functional performance: Habituel gait speed | Baseline, end of week 10
  Changes in habitual gait speed
Functional performance: Maximal gait speed | Baseline, end of week 10
  Changes in maximal gait speed
Functional performance: Sit-to-stand | Baseline, end of week 10
  Changes in sit-to-stand power.
Functional performance: Stair climb | Baseline, end of week 10
  Changes in stair climbing power
Resting metabolic rate | Baseline, end of week 10
  Changes in resting metabolic rate
Blood pressure: Systolic blood pressure | Baseline, end of week 10
  Changes in systolic blood pressure
Blood pressure: Diastolic blood pressure | Baseline, end of week 10
  Changes in diastolic blood pressure
Heart rate | Baseline, end of week 10
  Changes in resting heart rate
1 and 2-years cancer-specific survival | Randomization to 1 and 2 years after randomization
  Proportion of patients who have not died from gastroesophageal cancer 1 and 2 years after randomization
1 and 2-years over-all survival | Randomization to 1 and 2 years after randomization
  Proportion of patients who have not died 1 and 2 years after randomization
Progression-free survival | Randomization to 2 years after randomization
  Time to progression
Treatment tolerance: Hospitalization | 3, 6 and 9 weeks after randomization
  Unscheduled hospitalization
Treatment tolerance: Relative dose intensity | 3, 6 and 9 weeks after randomization
  Treatment tolerance assessed by the delivery of chemotherapy (relative dose intensity)
Treatment tolerance: Number of series recieved | 3, 6 and 9 weeks after randomization
  Treatment tolerance assessed by the delivery of chemotherapy (number of series recieved)
Treatment tolerance: Tolerated dose | 3, 6 and 9 weeks after randomization
  Treatment tolerance assessed by the delivery of chemotherapy (dose reduction)
Treatment tolerance: Permanent discontinuation of the treatment | 3, 6 and 9 weeks after randomization
  Treatment tolerance assessed by the delivery of chemotherapy (permanent discontinuation of the treatment)
Treatment effect: Response to chemotherapy | Randomization to 2 years after randomization
  Response to chemotherapy assessed by Response Evaluation Criteria in Solid Tumors 1.1 (complete response, partiel response, stable disease, progressive disease)
Health-related quality of life: Physical well-being | Baseline, 10 weeks-, 1 year-, and 2 years after randomization
  Changes in patient-reported physical well-being assessed using the Functional Assessment of Cancer Therapy - Esophagus (FACT-E) (scale-scoring 0-28, the higher the score the better quality of life)
Health-related quality of life: Social well-being | Baseline, 10 weeks-, 1 year-, and 2 years after randomization
  Changes in patient-reported social well-being assessed using FACT-E (scale-scoring 0-28, the higher the score the better quality of life)
Health-related quality of life: Emotional well-being | Baseline, 10 weeks-, 1 year-, and 2 years after randomization
  Changes in patient-reported social well-being assessed using FACT-E (scale-scoring 0-24, the higher the score the better quality of life)
Health-related quality of life: Functional well-being | Baseline,10 weeks-, 1 year-, 2 years after randomization
  Changes in patient-reported functional well-being assessed using FACT-E (scale-scoring 0-28, the higher the score the better quality of life)
Health-related quality of life: gastroesophageal cancer specific | Baseline, 10 weeks-, 1 year-, and 2 years after randomization
  Changes in patient-reported gastroesophageal cancer specific well-being assessed using FACT-E (scale-scoring 0-68, the higher the score the better quality of life)
Health-related quality of life: cancer cachexia specific | Baseline, 10 weeks-, 1 year-, and 2 years after randomization
  Changes in patient-reported cancer cachexia specific well-being assessed using Functional Assessment of Cancer Therapy - Cancer Cachexia (scale-scoring 0-48, the higher the score the better quality of life)
Depression | Baseline, 10 weeks-, 1 year-, and 2 years after randomization
  Changes in patient-reported depression, assessed using the Hospital Anxiety and Depression Scale (HADS) (scale scoring: 0-21, the higher the score the worse the condition)
Anxiety | Baseline, 10 weeks-, 1 year-, and 2 years after randomization
  Changes in patient-reported anxiety, assessed using the HADS (scale scoring: 0-21, the higher the score the worse the condition)
Self-reported physical activity: Walking | Baseline, end of week 10
  Changes in patient-reported weekly duration of walking, assessed using the International Physical Activity Questionnaire (IPAQ)
Self-reported physical activity: Moderate intensity physical activity (PA) | Baseline, end of week 10
  Changes in patient-reported weekly duration of moderate intensity PA, assessed using the IPAQ
Self-reported physical activity: Vigorous intensity PA | Baseline, end of week 10
  Changes in patient-reported weekly duration of vigorous intensity PA, assessed using the IPAQ
Self-reported physical activity: Total PA | Baseline, end of week 10
  Changes in patient-reported weekly duration of total PA, assessed using the IPAQ (Expressed as metabolic equivalent (MET)-min per week: MET level x minutes of activity x events per week)
Self-reported physical activity: Sitting time | Baseline, end of week 10
  Changes in patient-reported weekly duration of sitting time, assessed using the IPAQ
Self-reported screening of sarcopenia | Baseline, end of week 10
  Changes in patient-reported signs of sarcopenia, assessed using The Strength, assistance in walking, rise from a chair, climb stairs, and falls (SARC-F) questionnaire (scale scoring: 0-10, the higher the score the better the condition)
Self-reported three-days dietary records | Baseline, week 5 and week 10
  Changes in patient-reported three-day record of dietary intake assessed using questionnaries.
Patient-reported symptomatic adverse events | One week after each serie of chemotherapy during the intervention (10 weeks)
  Patient-reported symptomatic adverse events, assessed using the using the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)

OTHER OUTCOMES:
Blood biochemistry: Leukocyte differential counts | Baseline, end of week 10
  Changes in differential counts (total and per type: eosinofils, basofils, neutrofils, monocytes and lymphocytes)
Blood biochemistry: C-reactive protein | Baseline, end of week 10
  Changes in C-reactive protein
Blood biochemistry: albumin and protein | Baseline, end of week 10
  Changes in albumine and protein
Blood biochemistry: magnesium and phosphate | Baseline, end of week 10
  Changes in magnesium and phosphate
Blood biochemistry: Total cholesterol | Baseline, end of week 10
  Changes in total cholesterol
Blood biochemistry: Low-density lipoprotein cholesterol | Baseline, end of week 10
  Changes in low-density lipoprotein cholesterol
Blood biochemistry: High-density lipoprotein cholesterol | Baseline, end of week 10
  Changes in high-density lipoprotein cholesterol
Blood biochemistry: Triglyceride | Baseline, end of week 10
  Changes in triglyceride
Blood biochemistry: Glycated hemoglobin A1c | Baseline, end of week 10
  Changes in glycated hemoglobin A1c
Blood biochemistry: Insulin | Baseline, end of week 10
  Changes in insulin
Blood biochemistry: Glucose tolerance | Baseline, end of week 10
  Changes in glucose tolerance (2-hpur oral glucose tolerance test)
Blood biochemistry: Glucose | Baseline, end of week 10
  Changes in glucose
Blood biochemistry: C-peptide | Baseline, end of week 10
  Changes in c-peptide
Blood biochemistry: Interleukin-1 | Baseline, end of week 10
  Changes in interlieukin-1
Blood biochemistry: Interleukin-6 | Baseline, end of week 10
  Changes in interlieukin-6
Blood biochemistry: Interleukin-8 | Baseline, end of week 10
  Changes in interlieukin-8
Blood biochemistry: Interleukin-10 | Baseline, end of week 10
  Changes in interlieukin-10
Blood biochemistry: Interferon-gamma | Baseline, end of week 10
  Changes in interferon-gamma
Blood biochemistry: Tumor necrosis factor-alpha | Baseline, end of week 10
  Changes in tumor necrosis factor-alpha
Blood biochemistry: Circulating tumor DNA | Baseline, week 5 and 10
  Changes in circulating tumor DNA
Effect of acute exercise: Insulin sensitivity | Immediately after acute exercise
  Muscle glucose uptake during insulin stimulation after acute exercise
Effect of acute exercise: muscle protein synthesis | Immediately after acute exercise
  Muscle protein synthesis during insulin stimulation after acute exercise.
Changes of proteins in muscle biopsies | Before and immediately after acute exercise
  Modifications of proteins after acute exercise. Muscle biopsies will be subjected to mass spectrometry-based proteomic analysis.
Changes of proteins in mithocondrial regulation | Before and immediately after acute exercise
  Modifications of mithochondrial regulation. Signaling of mitochondiral fission, fusion and mitophagy will be examined in mucle biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Casper Simonsen, PhD, Principal Investigator — Copenhagen University Hospital, Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No